CLINICAL TRIAL: NCT03378752
Title: Atelectasis Formation Using High Frequency Jet Ventilation During Stereotactic Solid Organ Ablations
Brief Title: Atelectasis Formation Using HFJV During Stereotactic Solid Organ Ablations
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Jacob Freedman, Senior Consultant, Associate Professor, Karolinska Institutet
Other Study IDs: 2017/1158-32
Record Dates: First submitted 2017-12-04; First posted 2017-12-20 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: High Frequency Jet Ventilation; Atelectasis
Keywords: Computer tomography; Liver tumor thermoablation
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Atelectasis formation using HFJV: Computed tomography scans are performed every 15 minute during the first 45 minutes during general anaesthesia using high frequency jet ventilation.
  Interventions: Procedure: HFJV

INTERVENTIONS:
Procedure: HFJV — On High frequency jet ventilation, Every 15 minutes, after induction of general anaesthesia, a computed tomography of the lower part of the lungs are taken (10 cm volume, with the top of the right diaphragm as the lower border)

SUMMARY:
Atelectasis formation using HFJV during stereotactic solid organ ablations.

Primary endpoint will be to study the formation of atelectasis during HFJV. Secondary endpoint will be to study liver displacement over time. Reference groups will be found in previous published articles as referred to above.

Materials and methods: A radiological protocol has been made for the CT-scanner to take 10 cm volume Scans of the lower part of the lung. The scans will have its' lower border tangential to the top of the diaphragm. The first scan will be performed in the same session as the routine scan of the liver is performed after the patient is anesthetized. These Scans will then be repeated every 15 minute during the first 45 minutes. Arterial bloodgas analysis, transcutaneous CO2, blood pressure, saturation as well as parameters from the jet ventilator and the standard ventilator will be recorded.

DETAILED DESCRIPTION:
The use of HFJV in abdominal surgery as well as in out-of-operating theatre environment, is not well studied. In percutaneous liver thermal ablation the patient is anesthetized and intubated on the CT-bed where the liver ablation procedure is performed. Atelectasis is formed as soon as the patient is supine. Anesthesia itself also contributes to this. In extreme cases almost half the lung can be collapsed during anaesthesia, before any surgery has taken place.

The investigators have noticed that during this specific surgery, dynamic lung compliance does not necessarily worsen during HFJV but rather being unchanged or in some cases even becoming better and want to study this further and investigate the formation of atelectasis during HFJV. There are studies where atelectasis has been measured in a similar way as in this planned study, that is, with thin axial CT-scans at representative levels of the lung. This is during conventional lung ventilation, and has not yet been studied during HFJV.

Inclusion criteria: A total of n= 25 patients planned for elective liver tumor thermal ablation will be recruited after written informed consent.

Exclusion criteria: Patients 1/ under the age of 50 years, 2/with severe, poorly controlled lung disease.

The lung images will be saved in DICOM format and the tissue density will be analysed quantitatively. For each scan, the inner contour of each hemithorax will be manually drawn, excluding the chest wall, mediastinum, pleural effusions, and regions representing partial volume effects. Liver displacement can be measured from the routine CT-scans taken before and after the procedure.

Statistical methods: Chi2-analysis will be used to calculate the percentage of atelectasis in the lung.

Power calculation: Since the rate of atelectasis formation in the study groups is not known, it is impossible to perform power calculation for this trial. This study may clarify this issue in the planning of further studies.

This study may contribute to more knowledge about HFJV and its' effect on lung physiology, it may also contribute as a generator of new hypothesis and it might be a follow up study where the effect of alveolar recruitment maneuver (ARM) is studied.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients admitted to and by the surgeon planned for liver thermal ablation with cascination navigation system (requiring high frequency jet ventilation) from start date 25th of October, until a total number of 25 patients are included.

Exclusion Criteria:

* Age < 50 years old. Severe lung disease.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients referred for computed tomography guided ablation of liver tumours.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2017-12-19 (Actual); Study Completion 2017-12-19 (Actual)

PRIMARY OUTCOMES:
Change in formation of atelectasis during high frequency jet ventilation | Time frame is during surgery.
  Computed tomography Scans will be taken during general anaesthesia at the start of jet ventilation, t=0, and then at t=15 minutes, t=30 minutes and t=45 minutes. A total number of four scans will be performed in each study subject.

SECONDARY OUTCOMES:
Change of liver displacement | Time frame is during surgery.
  Routine CT Scans taken during surgery will be studied to calculate liver displacement over time.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institute Danderyd Hospital, Stockholm, Sweden

REFERENCES:
- [Background] Reinius H, Jonsson L, Gustafsson S, Sundbom M, Duvernoy O, Pelosi P, Hedenstierna G, Freden F. Prevention of atelectasis in morbidly obese patients during general anesthesia and paralysis: a computerized tomography study. Anesthesiology. 2009 Nov;111(5):979-87. doi: 10.1097/ALN.0b013e3181b87edb. PMID 19809292
- [Background] Denys A, Lachenal Y, Duran R, Chollet-Rivier M, Bize P. Use of high-frequency jet ventilation for percutaneous tumor ablation. Cardiovasc Intervent Radiol. 2014 Feb;37(1):140-6. doi: 10.1007/s00270-013-0620-4. Epub 2013 May 2. PMID 23636246
- [Background] Magnusson L, Spahn DR. New concepts of atelectasis during general anaesthesia. Br J Anaesth. 2003 Jul;91(1):61-72. doi: 10.1093/bja/aeg085. No abstract available. PMID 12821566
- [Background] Abderhalden S, Biro P, Hechelhammer L, Pfiffner R, Pfammatter T. CT-guided navigation of percutaneous hepatic and renal radiofrequency ablation under high-frequency jet ventilation: feasibility study. J Vasc Interv Radiol. 2011 Sep;22(9):1275-8. doi: 10.1016/j.jvir.2011.04.013. Epub 2011 Jun 23. PMID 21703873